CLINICAL TRIAL: NCT00240981
Title: Testosterone Replacement for Older Men With Sarcopenia
Brief Title: TOM: Testosterone in Older Men With Sarcopenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Higher incidence of cardiovascular events in the testosterone arm of the trial. Decision taken by the DSMB on December 31st, 2009.
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shalender Bhasin, Professor of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG0057; U01AG014369 (NIH)
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Sarcopenia; Hypogonadism; Muscular Diseases
Keywords: Andropause; frailty; hormone replacement therapy; Aging
MeSH Terms: conditions — Sarcopenia; Hypogonadism; Muscular Diseases; Frailty | interventions — Testosterone; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Topical testosterone gel 1% (active formulation)
- Placebo (Placebo Comparator)
  Interventions: Drug: Topical gel (placebo formulation)

INTERVENTIONS:
Drug: Topical testosterone gel 1% (active formulation) — Starting dose 10 g/day; increased to 15 g/day or decreased to 5 g/day in order to attain morning total testosterone level between 500 - 1000 ng/dL. Blinding achieved by combining a total of 3 tubes of active or placebo gel, applied to upper arms and shoulders each day.
  Other Names: Testim®
  Arms: Treatment
Drug: Topical gel (placebo formulation) — Starting dose 15 g/day (3 tubes), applied to upper arms and shoulders each day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether testosterone replacement in older men with low testosterone levels will increase muscle strength, improve physical performance and overall sense of well being, and reduce fatigue.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether testosterone replacement in older men, who have low testosterone levels and mild to moderate physical impairment, will increase their maximal voluntary muscle strength of major upper and lower extremity muscle groups. The second objective is to determine whether testosterone replacement will improve the power of knee extension, physical performance tests, the level of physical activity (measured by 3D accelerometer), self-reported disability, exercise tolerance and mobility. The third objective is to determine whether testosterone supplementation improves fatigue, affect, and overall sense of well being in older men with low testosterone levels. A fourth objective is to define the Minimum Clinically Important Differences in physical measures perceived by the participants (MCID).

Participant involvement will require 15-17 clinic visits over 28 weeks. Five to 7 of these visits are for physical testing, including body composition, muscle performance, and physical function. Throughout the study, hormone measurements will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling, ages 65 and older
* Self-reported difficulty in climbing 10 steps without resting, or difficulty in walking 2 or 3 blocks outside on level ground
* A score of 4 to 9 on the Short Physical Performance Battery (mild to moderate physical impairment)
* Total serum testosterone level (TT) < 350 ng/dL and > 100 ng/dL
* Without dementia (Mini-Mental State Examination [MMSE] score > 24)

Exclusion Criteria:

* Use of testosterone, anabolic steroids, dehydroepiandrosterone (DHEA), androstenedione or recombinant growth hormone (rGH) in the past year
* Alcohol or drug abuse
* Use of anti-convulsants or glucocorticoids (equivalent to prednisone > 20 mg/day)
* Prostate cancer, breast cancer or other cancers with life expectancy < 5 years
* Limiting neuromuscular, joint or bone disease, or history of stroke with residual neurological problems
* Any neurological condition that would impact cognitive functioning including:

  * epilepsy
  * multiple sclerosis
  * HIV
  * Parkinson's disease
  * stroke
  * other focal lesion
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) Axis I psychiatric disorder in past year or use of psychotropic medications in 6 months
* Abnormal prostate examination; PSA > 4 ng/mL; or BPH symptom score > 21
* Unstable angina, New York (NY) class III or IV congestive heart failure or myocardial infarction within 3 months of entry
* Abnormal laboratory values (at discretion of principal investigator)
* Untreated thyroid disease; systolic blood pressure > 160 or diastolic > 100 mm Hg
* Body mass index > 40 kg/m2
* Untreated severe obstructive sleep apnea

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 209 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Boston University Medical Center, Section of Endocrinology, Diabetes, and Nutrition; Shehzad Basaria, MD, Study Director — Boston University Medical Center, Section of Endocrinology, Diabetes, and Nutrition; Wildon Farwell, MD, MPH, Principal Investigator — VA Boston Healthcare System (Jamaica Plain Campus)
Locations (2):
- United States (2):
  - Boston University Medical Center, Boston, Massachusetts
  - VA Boston Healthcare System (Jamaica Plain Campus), Boston, Massachusetts

REFERENCES:
- [Background] Hughes VA, Frontera WR, Roubenoff R, Evans WJ, Singh MA. Longitudinal changes in body composition in older men and women: role of body weight change and physical activity. Am J Clin Nutr. 2002 Aug;76(2):473-81. doi: 10.1093/ajcn/76.2.473. PMID 12145025
- [Background] Hughes VA, Frontera WR, Wood M, Evans WJ, Dallal GE, Roubenoff R, Fiatarone Singh MA. Longitudinal muscle strength changes in older adults: influence of muscle mass, physical activity, and health. J Gerontol A Biol Sci Med Sci. 2001 May;56(5):B209-17. doi: 10.1093/gerona/56.5.b209. PMID 11320101
- [Background] Harman SM, Metter EJ, Tobin JD, Pearson J, Blackman MR; Baltimore Longitudinal Study of Aging. Longitudinal effects of aging on serum total and free testosterone levels in healthy men. Baltimore Longitudinal Study of Aging. J Clin Endocrinol Metab. 2001 Feb;86(2):724-31. doi: 10.1210/jcem.86.2.7219. PMID 11158037
- [Background] Gray A, Berlin JA, McKinlay JB, Longcope C. An examination of research design effects on the association of testosterone and male aging: results of a meta-analysis. J Clin Epidemiol. 1991;44(7):671-84. doi: 10.1016/0895-4356(91)90028-8. PMID 1829756
- [Result] Basaria S, Coviello AD, Travison TG, Storer TW, Farwell WR, Jette AM, Eder R, Tennstedt S, Ulloor J, Zhang A, Choong K, Lakshman KM, Mazer NA, Miciek R, Krasnoff J, Elmi A, Knapp PE, Brooks B, Appleman E, Aggarwal S, Bhasin G, Hede-Brierley L, Bhatia A, Collins L, LeBrasseur N, Fiore LD, Bhasin S. Adverse events associated with testosterone administration. N Engl J Med. 2010 Jul 8;363(2):109-22. doi: 10.1056/NEJMoa1000485. Epub 2010 Jun 30. PMID 20592293
- [Derived] Lee H, Hwang EC, Oh CK, Lee S, Yu HS, Lim JS, Kim HW, Walsh T, Kim MH, Jung JH, Dahm P. Testosterone replacement in men with sexual dysfunction. Cochrane Database Syst Rev. 2024 Jan 15;1(1):CD013071. doi: 10.1002/14651858.CD013071.pub2. PMID 38224135
- [Derived] Traustadottir T, Harman SM, Tsitouras P, Pencina KM, Li Z, Travison TG, Eder R, Miciek R, McKinnon J, Woodbury E, Basaria S, Bhasin S, Storer TW. Long-Term Testosterone Supplementation in Older Men Attenuates Age-Related Decline in Aerobic Capacity. J Clin Endocrinol Metab. 2018 Aug 1;103(8):2861-2869. doi: 10.1210/jc.2017-01902. PMID 29846604
- [Derived] Bhasin S, Travison TG, O'Brien L, MacKrell J, Krishnan V, Ouyang H, Pencina K, Basaria S. Contributors to the substantial variation in on-treatment testosterone levels in men receiving transdermal testosterone gels in randomized trials. Andrology. 2018 Jan;6(1):151-157. doi: 10.1111/andr.12428. Epub 2017 Oct 5. PMID 28981994
- [Derived] Gagliano-Juca T, Storer TW, Pencina KM, Travison TG, Li Z, Huang G, Hettwer S, Dahinden P, Bhasin S, Basaria S. Testosterone does not affect agrin cleavage in mobility-limited older men despite improvement in physical function. Andrology. 2018 Jan;6(1):29-36. doi: 10.1111/andr.12424. Epub 2017 Sep 26. PMID 28950424
- [Derived] Huang G, Bhasin S, Tang ER, Aakil A, Anderson SW, Jara H, Davda M, Travison TG, Basaria S. Effect of testosterone administration on liver fat in older men with mobility limitation: results from a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2013 Aug;68(8):954-9. doi: 10.1093/gerona/gls259. Epub 2013 Jan 4. PMID 23292288
- [Derived] Travison TG, Basaria S, Storer TW, Jette AM, Miciek R, Farwell WR, Choong K, Lakshman K, Mazer NA, Coviello AD, Knapp PE, Ulloor J, Zhang A, Brooks B, Nguyen AH, Eder R, LeBrasseur N, Elmi A, Appleman E, Hede-Brierley L, Bhasin G, Bhatia A, Lazzari A, Davis S, Ni P, Collins L, Bhasin S. Clinical meaningfulness of the changes in muscle performance and physical function associated with testosterone administration in older men with mobility limitation. J Gerontol A Biol Sci Med Sci. 2011 Oct;66(10):1090-9. doi: 10.1093/gerona/glr100. Epub 2011 Jun 22. PMID 21697501
- [Derived] LeBrasseur NK, Lajevardi N, Miciek R, Mazer N, Storer TW, Bhasin S. Effects of testosterone therapy on muscle performance and physical function in older men with mobility limitations (The TOM Trial): design and methods. Contemp Clin Trials. 2009 Mar;30(2):133-40. doi: 10.1016/j.cct.2008.10.005. Epub 2008 Oct 29. PMID 18996225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants provided written, informed consent. Recruitment took place at VAHCS, NERI, and BUMC. Outcome assessments were performed at BUMC. The study consisted of a 24- week intervention followed by a 12-week observation period. Enrollment took place between September 2005 and December 2009.
Pre-assignment Details: The participants were community-dwelling men, aged 65 years and older, with total testosterone between 100 and 350 ng/dL or free testosterone less than 50 pg/mL, and mobility limitation.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 106 | 103
Intent to Treat Sample | 82 | 83
Completed | 68 | 70
Not Completed | 38 | 33

BASELINE CHARACTERISTICS:
Population: Community-dwelling men, 65 years of age or older, with limitations in mobility and a total serum testosterone level of 100 to 350 ng per deciliter or a free serum testosterone level of less than 50 pg per milliliter were randomly assigned to receive placebo gel or testosterone gel, to be applied daily for 6 months.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 106 | 103 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 106 | 103 | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74 (6) | 74 (5) | 74 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 106 | 103 | 209
Region of Enrollment [Number; unit: participants]
  United States | 106 | 103 | 209

OUTCOME MEASURES:

1. Primary Outcome: Changes in Physical Performance Measured by an Exercise Testing Regimen
Description: Primary outcome was a change from baseline in leg-press strength at 6 months.
Time Frame: baseline and 6 months
Population: Participants with baseline and at least one post baseline measure.
Measure: Mean (95% Confidence Interval); unit: Newtons
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 49 | 54
Newtons | 156.9 [89.2 to 224.6] | 27.1 [-28.3 to 82.6]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — The unadjusted analysis using two-sample Student's t-tests of equal change in the trial groups, allowing unequal variance; Mean Difference (Net) = 129.8, 95% CI 2-sided [43.9 to 215.6]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.004, Regression, Linear — Adjusted analysis used multiple linear regression, with adjustment for baseline total score on the Short Physical Performance Battery, and self-report of limitations in mobility; Mean Difference (Net) = 129.4, 95% CI 2-sided [43.5 to 215.4]

2. Secondary Outcome: Chest-Press
Description: Change from baseline in chest press strength at 6 months
Time Frame: baseline and 6 months
Population: Participants with baseline and 1 post baseline measure.
Measure: Mean (95% Confidence Interval); unit: Newtons
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 38 | 44
Newtons | 34.7 [18.7 to 51.4] | 0.28 [-13.8 to 14.3]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — Unadjusted; Mean Difference (Net) = 34.5, 95% CI 2-sided [13.2 to 55.8]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Linear — Adjusted; Mean Difference (Net) = 34.5, 95% CI 2-sided [13.1 to 56.2]

3. Secondary Outcome: Stair-climbing Test (Without a Load)
Description: Change from baseline in the stair-climbing test (without a load) at 6 months.
Time Frame: baseline and 6 month
Population: Participants with baseline and one post baseline measure.
Measure: Mean (95% Confidence Interval); unit: Watts
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 49 | 52
Watts | 19.5 [7.4 to 31.5] | 10.7 [-2.9 to 24.3]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.34, t-test, 2 sided — Unadjusted; Mean Difference (Net) = 8.7, 95% CI 2-sided [-9.2 to 26.7]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.37, Regression, Linear — Adjusted; Mean Difference (Net) = 8.1, 95% CI 2-sided [-9.9 to 26.2]

4. Secondary Outcome: Grip Strength
Description: Change from baseline in grip strength in the dominant hand.
Time Frame: baseline and 6 months
Population: The participants with baseline and one post baseline measure are included.
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 63 | 70
Kilograms | 1.0 [-0.1 to 2.0] | 0.7 [-0.3 to 1.7]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.69, t-test, 2 sided — Unadjusted; Mean Difference (Net) = .27, 95% CI 2-sided [-1.1 to 1.7]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.71, Regression, Linear — Adjusted; Mean Difference (Net) = 0.26, 95% CI 2-sided [-1.1 to 1.7]

5. Secondary Outcome: 50-Meter Walking Speed (Without a Load)
Description: Change from baseline 50-Meter Walking Speed (without a load) at 6 months
Time Frame: baseline and 6 months
Population: Participants with a baseline and one post baseline measure.
Measure: Mean (95% Confidence Interval); unit: meters/second
Groups:
- Testosterone: Topical testosterone gel 1% (active formulation): Starting dose 10 g/day; increased to 15 g/day or decreased to 5 g/day in order to attain morning total testosterone level between 500 - 1000 ng/dL. Blinding achieved by combining a total of 3 tubes of active or placebo gel, applied to upper arms and shoulders each day.
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 39 | 43
meters/second | 0.074 [-0.004 to 0.153] | 0.024 [-0.018 to 0.066]
Statistical Analysis 1: Comparison: Testosterone vs Placebo; Test type: Superiority or Other; p = 0.26, t-test, 2 sided — Unadjusted; Mean Difference (Net) = 0.050, 95% CI 2-sided [-0.035 to 0.135]
Statistical Analysis 2: Comparison: Testosterone vs Placebo; Test type: Superiority or Other; p = 0.27, Regression, Linear — Adjusted; Mean Difference (Net) = 0.048, 95% CI 2-sided [-0.037 to 0.133]

6. Secondary Outcome: Stair-climbing Test (Loaded)
Description: Change from baseline in Stair-climbing Test (loaded)
Time Frame: baseline and 6 months
Population: Participants with one baseline and one post baseline measure.
Measure: Mean (95% Confidence Interval); unit: Watts
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 46 | 50
Watts | 39.2 [14.4 to 64.0] | 9.0 [-8.4 to 26.4]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — Unadjusted; Mean Difference (Net) = 30.2, 95% CI 2-sided [0.3 to 60.1]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.05, Regression, Linear — Adjusted; Mean Difference (Net) = 29.7, 95% CI 2-sided [0.2 to 59.3]

7. Secondary Outcome: Late Life Functional Disability Index (LLFDI)
Description: Percent change from baseline in the late life functional disability index at 6 months
Time Frame: baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 56 | 55
units on a scale | 61.2 [38 to 100] | 61.7 [38 to 100]

8. Secondary Outcome: Total Lean Mass
Time Frame: baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 82 | 81
Kilograms
  Baseline | 55.1 (6.9) | 56.5 (6.5)
  3 Months (N=73,75) | 57.2 (7.1) | 56.7 (6.2)
  6 Months (N=77,80) | 56.1 (6.9) | 56.2 (6.3)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.2, t-test, 2 sided — Month 3 Measures; Mean Difference (Net) = 1.8, 95% CI 2-sided [1.2 to 2.5]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p < .0001, t-test, 2 sided — Month 6 Measures; Mean Difference (Net) = 1.5, 95% CI 2-sided [0.4 to 2.2]

9. Secondary Outcome: Total Fat Mass
Time Frame: baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 82 | 81
Kilograms
  Baseline (N=82,81) | 26.2 (7.5) | 28 (8.4)
  3 Months (N=73,75) | 24.9 (7.1) | 28 (8.1)
  6 Months (N=77,80) | 24.0 (6.8) | 27.5 (7.9)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided — 3 Months Measures; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.7 to -0.6]
Statistical Analysis 2: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p < .0001, t-test, 2 sided — 6 Month Measures; Mean Difference (Net) = -2.0, 95% CI 2-sided [-2.8 to -1.2]

10. Secondary Outcome: 50-Meter Walking Speed (With a Load)
Description: Change from baseline 50-Meter Walking Speed (with a load) at 6 months
Time Frame: baseline and 6 months
Population: Participants with a baseline and one post baseline measure.
Measure: Mean (95% Confidence Interval); unit: meters/second
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 26 | 29
meters/second | 0.139 [0.023 to 0.256] | 0.065 [0.013 to 0.116]
Statistical Analysis 1: Comparison: Testosterone vs Placebo; Test type: Superiority or Other; p = 0.24, t-test, 2 sided — Unadjusted; Mean Difference (Net) = 0.074, 95% CI 2-sided [-0.05 to 0.19]
Statistical Analysis 2: Comparison: Testosterone vs Placebo; Test type: Superiority or Other; p = 0.14, Regression, Linear — Adjusted; Mean Difference (Net) = 0.090, 95% CI 2-sided [-0.030 to 0.209]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entire study period (4 years and 3 months)
Arm/Group | Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 16/106 | 8/103
Other Adverse Events (participants affected / at risk) | 35/106 | 10/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=106) | Placebo (N=103)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Diabetic foot ulcer (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Prostate cancer (Investigations) | 1 (1) | 0 (0)
Cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction treated with angioplasty, pacemaker placement (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Panic attack (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Angioplasty and coronary artery bypass grafting (Surgical and medical procedures) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Fracture of the tibia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Death, suspected myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Bupropion toxicity (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral angioplasty and stenting (Surgical and medical procedures) | 1 (1) | 0 (0)
Clozapine toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Congestive heart failure exacerbation (Cardiac disorders) | 1 (1) | 0 (0)
Community acquired pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Syncope resulting in hospitalization (Nervous system disorders) | 0 (0) | 1 (1)
Painful neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transurethral resection of prostate (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inflammatory colonic mass related to Crohn's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal bleeding from Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=106) | Placebo (N=103)
General disorders and administration site conditions (General disorders) | 5 (5) | 0 (0)
Infections and infestations (Infections and infestations) | 5 (5) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (6)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes